CLINICAL TRIAL: NCT03993639
Title: A Phase II Clinical Trial of KRN125 to Mobilize Hematopoietic Stem Cells Into Peripheral Blood in Healthy Volunteers
Brief Title: KRN125 for Mobilization of Hematopoietic Stem Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 125-101
Record Dates: First submitted 2019-05-23; First posted 2019-06-21 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Peripheral Blood Stem Cell Transplantation
Keywords: Hematopoietic Stem Cells Mobilization; Healthy Volunteer (HV); filgrastim; allogenic hematopoetic stem cell transplantation
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Intervention Model Description: Phase II, single center, open label, non-control, dose setting study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KRN125 (Experimental): Single SC administration
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Pegfilgrastim — Single dose of SC administration

SUMMARY:
Data collection to evaluate safety and effect of hematopoietic stem cell mobilization into the peripheral blood after a single subcutaneous (SC) dose of KRN125(Pegfilgrastim)in healthy adults.

DETAILED DESCRIPTION:
KRN125 is administered as a single SC dose to the Day 1. The stem cell mobilization protocols will be monitored for safety and efficacy during the mobilization period.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects aged 20 to 55 years or younger at the submission of the written informed consent form
* Women weighing 40 kg or more and 80 kg or less and men weighing 45 kg or more and 80 kg or less at the time of the preliminary examination

Exclusion Criteria:

* Subjects with a current medical history or who have been judged to be inappropriate for the study (e.g., significant neurological, hepatic, renal, endocrine, cardiovascular, blood, gastrointestinal, respiratory, and metabolic diseases, malignancies, myeloproliferative disorder, or psychiatric disorders)
* Individuals with alcohol or drug dependence, or individuals who have not tested negative for all drugs of abuse in the preliminary test
* Subjects with a history or current history of drug allergy or symptomatic allergy
* .Active infection or history of recurrent infection- However, only patients who are HBsantibody-positive by hepatitis B vaccination and whose HBV-DNA is less than the lower limit of quantitation will be allowed to participate in this study.
* Subjects who used drugs within 2 weeks before administration of the investigational drug.
* Subjects who have had at least 200 mL of blood drawn within 3 months before administration of the investigational drug.
* Pregnant or lactating

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Achievement of >20 cells/μL positive for CD34 in peripheral blood from baseline to Day 7 | Baseline to Day 7

SECONDARY OUTCOMES:
• Period from baseline to first time peripheral blood CD34 positive cells >20 cells/μL | Baseline to Day 15 or through study completion, an average of 1 year
• Time from baseline to peak peripheral blood CD34 positive cells | Baseline to Day 15 or through study completion, an average of 1 year
• Achievement of >10 cells/μL positive for CD34 in peripheral blood from baseline to Day 7 | Baseline to Day 7
• Peripheral blood CD34 positive cell count | Baseline to Day 15 or through study completion, an average of 1 year
• Peripheral blood white blood cell count | Baseline to Day 15 or through study completion, an average of 1 year
• Peripheral blood neutrophil count | Baseline to Day 15 or through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goto H, Sugita J, Hasegawa Y, Hayasaka K, Sunagoya K, Hatase R, Nishida M, Ichihashi Y, Odera M, Senjo H, Yokoyama S, Ara T, Shiratori S, Endo T, Hino M, Maeda Y, Sawa M, Sato N, Teshima T. Efficacy and Safety of Single-dose Pegfilgrastim for CD34 + Cell Mobilization in Healthy Volunteers: A Phase 2 Study. Transplantation. 2024 Apr 1;108(4):996-1003. doi: 10.1097/TP.0000000000004880. Epub 2024 Mar 23. PMID 38012835